CLINICAL TRIAL: NCT05713526
Title: The Effect of Telehealth Service Provided to Pregnant Women About Childhood Vaccines on Vaccine Attitudes and Vaccination
Brief Title: The Effect of Telehealth Service About Childhood Vaccines on Vaccine Attitudes and Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gozde AKSUCU (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor-Investigator, Gozde AKSUCU, Research Assistant, University of Beykent
Organization: University of Beykent (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021/295
Record Dates: First submitted 2023-01-25; First posted 2023-02-06 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Vaccine Refusal; Vaccination
Keywords: Telehealth; Vaccine hesitation; Vaccine attitudes; Vaccination; Childhood immunization
MeSH Terms: conditions — Vaccination Refusal

STUDY DESIGN:
Intervention Model Description: Pretest-posttest with the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth group (Experimental): The group in which telehealth services for childhood vaccines will be implemented.
  Interventions: Behavioral: Telehealth service
- Control group (No Intervention): The group in which telehealth services for childhood vaccines will not be implemented.

INTERVENTIONS:
Behavioral: Telehealth service — Researchers will send educational materials (video and e-brochures) about childhood vaccinations to the participants' mobile phones at regular intervals, answer their questions over the phone and send reminder messages before the vaccination appointment.
  Arms: Telehealth group

SUMMARY:
The goal of this clinical trial is to test the effect of telehealth service provided to pregnant women about childhood vaccines on vaccine attitudes and vaccination.

The main questions it aims to answer are:

* Does telehealth service provided to pregnant women about childhood vaccines decrease the mean scores of the vaccine attitudes scale?
* Does telehealth service provided to pregnant women about childhood vaccines increase the vaccination?

In the intervention group, researchers will send educational materials (video and e-brochures) about childhood vaccinations to the participants' mobile phones at regular intervals, answer their questions over the phone and send reminder messages before the vaccination appointment.

In the control group, there will be no information or intervention about childhood vaccines by the researchers, and standard procedure will be followed.

Researchers will compare the intervention and control groups to see if there is a difference between vaccination attitudes and vaccination rates.

DETAILED DESCRIPTION:
Place and Time of Research; The research will be carried out at primary care clinics in Istanbul Beylikdüzü between August 2022 and March 2023.

Population and Sample of the Research; The research population will consist of individuals who were last trimester of pregnancy in primary care clinics in Istanbul Beylikdüzü. The study sample will consist of at least 156 individuals determined by power analysis. Individuals who met the inclusion criteria were randomly assigned to the experimental and control groups with a table of random numbers.

In this study, the scales will be applied as a pre-post test. It does not pose any problem that will endanger the physical and mental health of the participants. Data collection forms; introductory information form, vaccine attitudes scale, vaccine follow-up form, and follow-up chart. Data collection tools; vaccination information video, e-brochures, reminder messages, answering parent questions via instant message, smartphone.

Before starting the research, ethics committee approval was obtained from Istanbul University-Cerrahpaşa Social and Human Sciences Ethics Committee, and institutional permission was obtained from the Istanbul Provincial Health Directorate. Participants were included in the study voluntarily. Before starting the study, participants were called by phone and informed about the study, and verbal consent was obtained with the "Informed Voluntary Consent Form."

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Having the ability to understand, speak, read and write Turkish.
* The willingness of the primary care clinic staff to be cooperated to work
* Owning and using a smartphone
* Being in the last trimester of pregnancy
* Giving birth to the baby at a birth weight (≥ 2000 g) that will not affect the routine vaccination schedule

Exclusion Criteria:

* Have a miscarriage

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Since pregnancy is specific to women, the study will be conducted for women.
Enrollment: 183 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Vaccine attitudes (Vaccine Attitudes Scale) | Before the intervention
  The scale was developed by Wallece et al. in 2019. The Turkish validity and reliability study was carried out by Ceylan et al. in 2021. The scale consists of 11 items in a 3-point Likert type that measures parents' attitudes toward vaccines. The scale has five sub-dimensions consisting of "benefits of the vaccine", "past vaccination behavior", "efficacy and safety", "awareness of vaccine-preventable diseases" and "confidence". Each item is scored between 1 and 3 (agree=1, undecided=2, disagree=3). The total score on the scale ranges from 11 to 33. 11 points indicate that parents have a positive attitude toward the vaccine, while 33 points indicate a negative attitude. The scale does not have a breakpoint. As the score obtained from the scale increases, the parents' hesitance toward vaccination increases, and that is, they show a negative attitude towards vaccination. Cronbach's alpha coefficient was calculated by Ceylan (2021) as 0.66 to evaluate the scale's internal consistency.
Vaccine attitudes (Vaccine Attitudes Scale) | After the 6th month's vaccinations
  The scale was developed by Wallece et al. in 2019. The Turkish validity and reliability study was carried out by Ceylan et al. in 2021. The scale consists of 11 items in a 3-point Likert type that measures parents' attitudes toward vaccines. The scale has five sub-dimensions consisting of "benefits of the vaccine", "past vaccination behavior", "efficacy and safety", "awareness of vaccine-preventable diseases" and "confidence". Each item is scored between 1 and 3 (agree=1, undecided=2, disagree=3). The total score on the scale ranges from 11 to 33. 11 points indicate that parents have a positive attitude toward the vaccine, while 33 points indicate a negative attitude. The scale does not have a breakpoint. As the score obtained from the scale increases, the parents' hesitance toward vaccination increases, and that is, they show a negative attitude towards vaccination. Cronbach's alpha coefficient was calculated by Ceylan (2021) as 0.66 to evaluate the scale's internal consistency.
Vaccination | When the birth occurs
  Vaccination status on the day of the appointment
Vaccination | When the baby is at the end of the 1st month
  Vaccination status on the day of the appointment
Vaccination | When the baby is at the end of the 2nd month
  Vaccination status on the day of the appointment
Vaccination | When the baby is at the end of the 4th month
  Vaccination status on the day of the appointment
Vaccination | When the baby is at the end of the 6th month
  Vaccination status on the day of the appointment

CONTACTS AND LOCATIONS:
Overall Officials: Gözde AKSUCU, MSc, Study Chair — Beykent University; Seda ÇAĞLAR, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Primary Care Clinics, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aksucu G, Caglar S. Effects of telehealth during pregnancy on childhood vaccine attitudes and timeliness: A randomized controlled trial. Vaccine. 2025 Sep 17;63:127678. doi: 10.1016/j.vaccine.2025.127678. Epub 2025 Aug 28. PMID 40882266